CLINICAL TRIAL: NCT02712216
Title: Evaluation of Abdominal Wall Thickness at Possible Trocar Sites Based on Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Lutz, Assistant Professor Obstetrics-Gynecology, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0298
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Surgery
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trocar Insertion Sites (Other): Insertion of a 21-gauge 3.5inch spinal needle perpendicular to the abdominal wall at each possible trocar site. The needle will be placed after the abdomen is insufflated under direct visualization with the laparoscopic camera. The needle will be inserted to the level of the peritoneum and a hemostat will be place on the needle at the level of the epidermis.
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Determine best port sites to insert bariatric trocars
  Other Names: Trocar Insertion Sites

SUMMARY:
The purpose of this research study is to determine which sites are best suited for laparoscopic entry of bariatric trocars in the morbidly obese population.

DETAILED DESCRIPTION:
Patients already scheduled for laparoscopy will be approached for participation prior to surgery. During laparoscopy, the investigators routinely inject port sites with a 21-gauge needle and inject sites with local anesthetic prior to trocar placement. In the study the investigators will insert a 21-gauge 3.5inch spinal needle perpendicular to the abdominal wall at each possible trocar site. The seven insertion sites are the umbilicus; 12cm lateral to umbilicus on right; 12cm lateral to umbilicus on left; Left lower quadrant lateral to inferior epigastric; Right lower quadrant lateral to inferior epigastric, Lower midline of abdomen; Left upper quadrant at Palmer's Point. The needle will be placed after the abdomen is insufflated under direct visualization with the laparoscopic camera. The needle will be inserted to the level of the peritoneum and a hemostat will be place on the needle at the level of the epidermis. The abdominal wall thickness will be measured with a ruler and recorded to the nearest millimeter. The information will be recorded on the case report form attached. The case report form will be kept in a binder in the research coordinators office.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-64; BMI greater than 18.5

Exclusion Criteria:

* Abdominal hernias

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Measurement of abdominal wall depths | Measurement of abdominal wall depth will occur during the surgical procedure
  The measurement will be evaluated based on the following BMI categories: BMI 18.5-24.9 (normal weight) BMI 25-29.9 (overweight) BMI 30-34.9 (class 1 obesity) BMI 35-39.9 (class 2 obesity) BMI >40 (class 3 obesity)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lutz, MD, Principal Investigator — University of Mississippi Medical Center
Locations (4):
- United States (4):
  - University Physician's Grant's Ferry, Flowood, Mississippi
  - University Physician's Women's Specialty Care, Flowood, Mississippi
  - University's Physician Specialty Clinics Jackson Medical Mall, Jackson, Mississippi
  - Winfred L. Wiser, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No